CLINICAL TRIAL: NCT02459119
Title: A Multicenter, Non-Randomized, Phase II Study of Regorafenib for Advanced Urothelial Cancer Following Prior Chemotherapy
Brief Title: Study of Regorafenib for Urothelial Cancer Following Chemotherapy (UAB 1477)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Principal Investigator, Lisle Nabell, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F150302002 (UAB 1477)
Record Dates: First submitted 2015-05-26; First posted 2015-06-01 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Urothelial Cancer (Urinary Bladder, Ureters, or Renal Pelvis Cancer)
Keywords: urothelial cancer; Regorafenib
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib (Experimental): Regorafenib will be administered orally to all patients on study. The drug will be taken once a day for 3 of every 4 week cycle (3 weeks on/1 week off). The dose is 120 mg once daily for the first cycle, then 160 mg once daily from the second cycle if no significant Regorafenib-associated toxicities occur during the first cycle. Drug dosage may be modified if toxicities occur. Patients will undergo up to 4 cycles of treatment and may continue on additional at the discretion of the investigator.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib will be packaged as 40 mg tablets in a bottle. Patients will be instructed to maintain a daily medication calendar.

SUMMARY:
This study will test how well Regorafenib controls disease progression in urothelial cancer (cancer occurring in the urinary bladder, ureters, or renal pelvis) following previous therapy with chemotherapy.

DETAILED DESCRIPTION:
Advanced urothelial carcinoma (UC) has a poor long-term prognosis. The disease has not seen improved outcomes despite research efforts in over two decades. Novel therapeutic options are needed. Regorafenib is a novel oral multikinase inhibitor but is more potent than a similar multikinase inhibitor drug that treats advanced renal cell carcinoma and hepatocellular carcinoma. Regorafenib has been shown to have a broader capacity to inhibit blood supply to tumor sources.

This trial evaluates a proof-of-concept using Regorafenib in patients with metastatic progressive urothelial carcinoma following chemotherapy but still have a high level of activity performance in their daily living. The initial dose of Regorafenib will be 120 mg daily and then be escalated to 160 mg daily before gradually tapering.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically proven transitional cell carcinoma of the urothelium.
* Progressive disease after 1-3 prior chemotherapy regimens (perioperative chemotherapy within 12 months will be considered one regimen).
* Prior regimen must be within 6 months of registration
* Measurable disease by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-1
* Patients with metastatic (lymph node or distant metastasis, i.e. N+ or M1) or locally advanced unresectable (T4b) transitional cell carcinoma.
* Age ≥19 years
* Life expectancy of at least 12 weeks (3 months)
* Subjects must be able to understand and be willing to sign the written informed consent form.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements:

  * Total bilirubin ≤ 1.5 x the upper limits of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
  * Alkaline phosphatase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
  * Serum creatinine ≤ 1.5 x the ULN
  * International normalized ratio (INR) less than or equal to 1.5 x ULN. (Subjects who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists.Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care.
  * Platelet count >100,000/mm3, hemoglobin (Hb) >8 g/dL, absolute neutrophil count (ANC) 1500/mm3. The patient cannot be transfused in order to meet study entry criteria.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post- menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test. The definition of adequate contraception will be based on the judgment of the investigator.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form until at least 3 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
* Subject must be able to swallow and retain oral medication.

Exclusion Criteria:

* Component of small-cell cancer or sarcomatoid cancer
* Prior therapy with any systemic therapy (chemotherapy or biologic therapy) within twenty-eight days prior to study entry
* Patients must have recovered from toxicities from prior systemic anticancer treatment or local therapies.
* Patients who have undergone major surgery <4 weeks or minor surgery <2 weeks prior to registration. Wounds must be completely healed prior to study entry and patients recovered from all toxicities from surgery. Placement of a vascular access device is not considered major or minor surgery in this regard.
* Prior radiation therapy is allowed as long as the irradiated area was not the sole source of measurable disease and radiotherapy was completed with recovery from toxicity, at least three weeks prior to enrollment. If the irradiated area is the only site of disease, there must be evidence of progressive disease.
* Uncontrolled central nervous system (CNS) metastases (previously treated with radiation and off steroids is acceptable).
* Patient with active or uncontrolled infection.
* Recent or active bleeding diathesis or arterial vascular event within 4 weeks.
* Pregnant or nursing (Fertile patients must use effective contraception during and for up to 3 months after completion of study treatment.)
* Patients may not be receiving any other investigational agents.
* Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter study.
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure >90 mm Hg on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) Class II.
  * Active coronary artery disease.
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
  * Unstable angina (angina symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment within 6 months of informed consent.
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from breast cancer except cervical cancer in-situ, treated localized basal cell carcinoma, Gleason score 6 prostate cancer or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before randomization are allowed. All cancer treatments for another malignancy must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form).
* Patients with pheochromocytoma.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Ongoing infection >Grade 2 NCI-CTCAE v4.0.
* Symptomatic metastatic brain or meningeal tumors.
* Presence of a non-healing wound, non-healing ulcer, or bone fracture.
* Renal failure requiring hemo-or peritoneal dialysis.
* Dehydration Grade >1 NCI-CTCAE v4.0.
* Patients with seizure disorder requiring medication.
* Persistent proteinuria greater than or equal to Grade 3 NCI-CTCAE v4.0 (> 3.5 g/24 hrs, measured by urine protein:creatinine ratio on a random urine sample).
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI- CTCAE version 4.0 Grade 2 dyspnea).
* History of organ allograft (including corneal transplant).
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
* Any malabsorption condition.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-05; Primary Completion 2019-02 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisle Nabell, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Wayne State University, Detroit, Michigan
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regorafenib
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants were treated and eligible for analysis
Arm/Group | Regorafenib
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 67.5 [55 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival at 6 Months
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Death is also considered as progression in the analysis.
Time Frame: Baseline to 6 months following start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 17
Participants | 3

2. Secondary Outcome: Disease Response Rate
Description: The number of participants showing response at first restaging scan after the start of study treatment. The response will be assessed using tumor measurements which will be documented through CT scans, magnetic resonance imaging (MRI), and x-rays using the Response Evaluation Criteria in Solid Tumors (RECIST). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: Every 8 weeks until the time of disease progression upto 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 17
Participants | 9

3. Secondary Outcome: Overall Survival
Description: Length of subject survival after starting study treatment
Time Frame: Baseline to 3 years
Measure: Mean (Standard Error); unit: days
Arm/Group | Regorafenib
Number analyzed (Participants) | 17
days | 100 (10.33)

4. Secondary Outcome: Rate of Progression-free Survival
Description: Duration of time from the start of treatment to time of progression or death, whichever comes first.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From start of treatment to time of progression or death, assessed up to 6 months
Measure: Mean (Standard Error); unit: days
Arm/Group | Regorafenib
Number analyzed (Participants) | 17
days | 47.6 (3.6)

5. Secondary Outcome: Number of Participants With Adverse Events
Description: The Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 will be used for assessment of toxicities.
Time Frame: At the end of first treatment until 6 months following last treatment, an expected average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 17
Participants | 13

ADVERSE EVENTS:
Time Frame: From the date of signing consent form until 6 months after stopping study treatment.
Arm/Group | Regorafenib
All-Cause Mortality (participants affected / at risk) | 8/17
Serious Adverse Events (participants affected / at risk) | 7/17
Other Adverse Events (participants affected / at risk) | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (N=17)
Anemia (Vascular disorders) | 1 (1) — Grade 3
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 3
Thrombocytopenia (Vascular disorders) | 1 (1) — Grade 3
Low Phospohorus (Musculoskeletal and connective tissue disorders) | 2 (2) — Grade 3
Fatigue (General disorders) | 1 (1) — Grade 3
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) — Grade 1 requiring intervention to prevent permanent damage
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (N=17)
Hand foot syndrome (Musculoskeletal and connective tissue disorders) | 3 (11) — None of them were grade 3 or higher
Hyponatremia (Vascular disorders) | 1 (1) — Grade 2
Hematuria (Vascular disorders) | 1 (1) — Grade 1
Dry eyes (Eye disorders) | 1 (1) — Grade 1
Diarrhea (Gastrointestinal disorders) | 2 (2) — Grade 1
Epistaxis (Vascular disorders) | 1 (1) — grade 1
Voice hoarseness (Ear and labyrinth disorders) | 1 (1) — Grade 1
Vomitting (Gastrointestinal disorders) | 1 (1) — Grade 2
intermittent tachycardia (Cardiac disorders) | 1 (1) — Grade 1
Hypomagnesemia (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT02459119/Prot_SAP_000.pdf